CLINICAL TRIAL: NCT05273723
Title: The Effect of a Multi-Component Behavior Change Technique Intervention on Physical Activity Among Individuals on Primary Prevention Statin Therapy: A Dose-Finding Pilot Study
Brief Title: A BCT Intervention for Physical Activity Among Individuals on Statins
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-0674; P30AG063786-01 (NIH)
Record Dates: First submitted 2021-12-27; First posted 2022-03-10 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Insufficient Physical Activity
Keywords: Behavior Change; Physical Activity; Walking; Statins; Cardiovascular Disease; Dose Finding; Continual Reassessment Method
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The study utilizes a modified Time-to-Event Continual Reassessment Method Dose-Finding Design
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Dose-finding study with 14 groups of 3 participants each. To identify the minimum effective dose (MED) to increase walking by 2,000 more steps per day between run-in and follow-up periods, the first group of 3 participants will receive a 5-week dose of the multi-BCT intervention. For the next subjects, the doses to administrate will vary between 1 and 10 weeks in length and will be determined using a modified version of the Time-to-Event Continual Reassessment Method (TiTE-CRM) according to the observed responses in the previous participants.
  Interventions: Behavioral: 5 Behavioral Change Techniques

INTERVENTIONS:
Behavioral: 5 Behavioral Change Techniques — 1. Goal setting: set or agree on a goal defined in terms of behavior to be achieved. Example: Set the goal of walking 2,000 steps more per day.
  2. Action planning: prompt detailed planning of performance of behavior (must include a setting [walking to the mailbox], frequency, duration, and intensity. Example: Develop a plan to walk today.
  3. Self-Monitoring of behavior: establish a method for person to monitor and record their number of steps based on their Fitbit. Example: Did you check your Fitbit and record daily total number of steps?
  4. Feedback on behavior: Monitor and provide informative or evaluative feedback on performance of the behavior (e.g. form, frequency, duration, intensity). Example: You walked 6,000 steps today.
  5. Prompts/Cues: introduce or define environmental or social stimulus with the purpose of prompting or cueing the behavior. The prompt or cue would normally occur at the time or place of performance. Example: You planned to walk today in the park at 3pm.

SUMMARY:
The purpose of this project is to identify the minimum effective dose (MED) of a multi-component behavioral change intervention required to increase levels of physical activity (PA) among participants on primary prevention statin therapy who are at elevated risk for cardiovascular disease (CVD). The intervention will be comprised of 5 BCTs which have previously shown to be effective on increasing health behaviors: Goal Setting, Action Planning, Self-Monitoring, Feedback, and Prompts/Cues. Participants will complete a 2-week baseline run-in period where PA levels will be measured using Fitbit wearable device. Then 42 participants will be randomized into 14 cohorts of 3 participants each for the intervention period. During the intervention period, participants will receive a multi-BCT intervention, the length of which varies between 1 and 10 weeks depending on the assigned dose. Assignment to doses will utilize a modified version of the Time-to-Event Continual Reassessment Method (TiTE-CRM) methodology to adjust the dose for each cohort based on the results from the previous cohort. After the intervention, there will be a 2-week follow-up period. The MED will be defined as the smallest BCT dose (defined by weeks of intervention) associated with 80% of participants having a successful PA increase between the run-in and the follow-up periods (defined as walking an extra 2,000 more steps per day).

DETAILED DESCRIPTION:
The purpose of this project is to identify the minimum effective dose (MED) of a multi-component behavioral change intervention required to increase levels of physical activity (PA) among participants on primary prevention statin therapy who are at elevated risk for cardiovascular disease (CVD). The long-term goal is to prevent CVD. The current project will utilize a modified version of the time-to-event continual reassessment method (TiTE-CRM), a state of the art dose finding methodology, to determine the MED of a multi-component behavioral change technique (BCT) intervention required to increase PA by an average of 2,000 steps per day. The intervention will be comprised of 5 BCTs which have previously shown to be effective on increasing health behaviors: Goal Setting, Action Planning, Self-Monitoring, Feedback, and Prompts/Cues.

The sample will include individuals on primary prevention statin therapy. For this research, the investigators will enroll currently sedentary persons, with the goal of randomizing 42 persons to the intervention. Enrolled participants will complete a 2-week run-in period where PA levels will be measured using Fitbit wearable devices and levels of adherence to statin medications will be assessed using a smart pill bottle. During the baseline run-in period, objective data from the Fitbit wearable devices will be used to verify sedentary behavior. Individuals who do not have objective levels of sedentary behavior and/or are non-adherent to the protocol will be excluded and will not be randomized to the intervention. Following run-in, the investigators will randomize 42 participants into 14 cohorts of 3 participants each for the intervention period. During the intervention period, participants will receive a multi-BCT intervention, the length of which varies between 1 and 10 weeks depending on the assigned dose. Assignment to doses will utilize modified TiTE-CRM methodology to adjust the dose for each cohort based on the results from the previous cohort. Following the intervention, all participants will be assessed over a 2-week follow-up period which includes passive data collection from the activity monitor, answering surveys, and use of smart pill bottle to track medication adherence. The MED will be defined as the smallest BCT dose duration associated with 80% of participants having a successful PA increase between the run-in and the follow-up periods. Change in PA will be defined as the difference in average daily PA between the run-in and follow-up periods. The investigators will also assess Mechanisms of Action (MoAs) to determine potential mediators of the BCT intervention on PA. As increasing PA may change statin adherence, the investigators will utilize smart pill bottle to measure adherence to statin medications.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older;
* Northwell Health employee/affiliate
* Ambulatory without limitations: has never been advised by a clinician that increasing low-intensity walking would be unsafe;
* Prescribed statin medication;
* Self-reported low levels of physical activity
* Access to and capable of using a smart cellular phone;
* After 2 week run-in, objectively-verified low levels of physical activity as documented by a commercially available Fitbit device
* English speaking.

Exclusion Criteria:

* Age less than 18 years;
* Not a Northwell Health employee/affiliate
* Non-ambulatory or unsafe/not recommended to participate in a walking program
* Not prescribed statin medication;
* History of CVD;
* Inability to comply with study protocol during 2 week run-in;
* Does not speak English;
* Unavailable for follow-up;
* Cognitive impairment;
* Severe mental illness (e.g., bipolar disorder or schizophrenia);
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Davidson, PhD, MASc, Principal Investigator — Northwell Health
Locations (1):
- Institute of Health System Science, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form following completion of recruitment but prior to publication of any data from the current study. De-identified, pooled individual participant data will be made available within a year of final participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
Access Criteria: All data and supporting information will be stored on the Open Science Framework, a free web application with no access restrictions.

REFERENCES:
- [Derived] Goodwin AM, Friel C, Miller D, Vicari F, Duer-Hefele J, Chandereng T, Davidson KW, Alfano CM, Cheung YK, Butler MJ. Minimum effective dose of a multicomponent behaviour change intervention to increase the physical activity of individuals on primary statin therapy: an adaptive study using the time-to-event continual reassessment method (TiTE-CRM). BMJ Open. 2025 Aug 5;15(8):e090789. doi: 10.1136/bmjopen-2024-090789. PMID 40764069
- [Derived] Butler MJ, Romain AN, Augustin R, Robles P, Friel CP, Vicari F, Chandereng T, Alfano CM, Cheung YK, Davidson KW. The effect of a multi-component behavior change technique intervention on physical activity among individuals on primary prevention statin therapy: A dose-finding trial protocol. Contemp Clin Trials. 2023 Jul;130:107205. doi: 10.1016/j.cct.2023.107205. Epub 2023 Apr 25. PMID 37105318

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The first two weeks of the study are a baseline assessment period. Participants will be mailed a commercially available Fitbit to wear day and night, and eCAP bottle to fill using their existing statin prescription. After successful completion of the baseline period, participants will move on to the intervention period.
Groups:
- Multi-BCT Intervention 5 Weeks: 5-week multi-component BCT intervention delivered via text messages
- Multi-BCT Intervention 6 Weeks: 6-week multi-component BCT intervention delivered via text messages
- Multi-BCT Intervention 8 Weeks: 8-week multi-component BCT intervention delivered via text messages
- Multi-BCT Intervention 9 Weeks: 9-week multi-component BCT intervention delivered via text messages
- Multi-BCT Intervention 10 Weeks: 10-week multi-component BCT intervention delivered via text messages
Period: Cohort 1: 5 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 3 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: 6 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 3 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 3: 8 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 4: 8 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 2 | 0 | 0
Completed | 0 | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 5: 9 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 6: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 7: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 8: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 9: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 10: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 11: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 12: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 13: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 14: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 15: 10 Week Intervention
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
Started | 0 | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 42 participants completed the 2-week baseline period
Groups:
- Intervention (All Participants): Dose-finding study with 13 groups of 3 participants each, 1 group of 2 participants, and 1 group of 1 participant. To identify the minimum effective dose (MED) to increase walking by 2,000 more steps per day between run-in and follow-up periods, the first group of 3 participants will receive a 5-week dose of the multi-BCT intervention. For the next subjects, the doses to administrate will vary between 1 and 10 weeks in length and will be determined using a modified version of the Time-to-Event Continual Reassessment Method (TiTE-CRM) according to the observed responses in the previous participants. Pre-specified to report results across the full sample.
Arm/Group | Intervention (All Participants)
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 29
  More than one race | 2
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a 2,000 Step/Day Increase Between run-in and Follow-up
Description: Participant steps will be assessed continuously using a Fitbit mobile device. Daily steps for participants will be aggregated by run-in and follow-up periods to generate average daily steps in each period. Average daily steps in the follow-up period will be compared to average daily steps in the run-in period. If the average steps in follow-up are 2,000 steps per day greater than during run-in, the outcome for the Time-to-Event Continual Reassessment Method (TiTE-CRM) will be judged successful. The minimum effective dose (MED) will be defined as the smallest BCT dose duration associated with 80% participants receiving that dose having a successful increase in walking between the run-in and the follow-up periods. Pre-specified to report primary and secondary outcome results across the full sample.
Time Frame: Mean daily step totals will be compared between the run-in (2 weeks pre-intervention) and follow-up periods (2 weeks post-variable intervention of 5-10 weeks).
Population: Results presented for the full sample. This is an adaptive trial using the TiTE-CRM. Doses are assigned using adaptive methods throughout the trial using all available data from all participants, regardless of enrollment cohort or dose assignment. As a result, there are no a priori hypotheses for comparing outcomes between dose levels. Of the 42 participants who received the intervention, 40 participants (95.2%) had sufficient data to generate estimates of the MED.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention (All Participants): To identify the minimum effective dose (MED) to increase walking by 2,000 more steps per day between run-in and follow-up periods, the first group of 3 participants will receive a 5-week dose of the multi-BCT intervention. For the next subjects, the doses to administrate will vary between 5 and 10 weeks in length and will be determined using a modified version of the Time-to-Event Continual Reassessment Method (TiTE-CRM) according to the observed responses in the previous participants. Pre-specified to report primary and secondary outcome results across the full sample.
Arm/Group | Intervention (All Participants)
Number analyzed (Participants) | 40
Participants | 7

2. Secondary Outcome: Within-person Change in Daily Steps.
Description: Participant steps will be assessed continuously using a Fitbit mobile device. Daily steps for participants will be aggregated by run-in and follow-up periods to generate average daily steps in each period. Changes in daily steps between run-in and intervention periods will be compared using Generalized Linear Mixed Model Analyses. Pre-specified to report primary and secondary outcome results across the full sample.
Time Frame: as for outcome 1
Population: Results presented for the full sample. This is an adaptive trial using the TiTE-CRM. Doses are assigned using adaptive methods throughout the trial using all available data from all participants, regardless of enrollment cohort or dose assignment. As a result, there are no a priori hypotheses for comparing outcomes between dose levels. Of the 42 participants who received the intervention, n=32 (76.2%) had sufficient data during the baseline and follow-up periods to include in analyses.
Measure: Mean (Standard Deviation); unit: steps/day
Groups:
- Intervention: To identify the minimum effective dose (MED) to increase walking by 2,000 more steps per day between run-in and follow-up periods, the first group of 3 participants will receive a 5-week dose of the multi-BCT intervention. For the next subjects, the doses to administrate will vary between 5 and 10 weeks in length and will be determined using a modified version of the Time-to-Event Continual Reassessment Method (TiTE-CRM) according to the observed responses in the previous participants. Pre-specified to report primary and secondary outcome results across the full sample.
Arm/Group | Intervention
Number analyzed (Participants) | 32
steps/day | -152.23 (2,596.99)

3. Secondary Outcome: Within-person Change in Self-Efficacy for Walking.
Description: Self-efficacy will be assessed using the Self-Efficacy for Walking (SE-W) scale, a 10-item measure assessing patient's capabilities to walk for durations of 5 to 50 minutes. Items are scored from 0 to 100%, with scores of 0% indicating participants are "not at all confident" they could walk for that duration and scores of 100% indicating the participants are "highly confident" they could walk that duration. Items are average to create a total score, with higher scores indicating higher levels of beliefs about self-efficacy. Pre-specified to report primary and secondary outcome results across the full sample.
Time Frame: Self-efficacy will be assessed at the completion of the 2-week run-in and at the end of the 2-week follow-up period. Changes in self-efficacy will be reported comparing mean difference scores between run-in and follow-up (follow-up mean minus run-in mean)
Population: Results presented for the full sample. This is an adaptive trial using the TiTE-CRM. Doses are assigned using adaptive methods throughout the trial using all available data from all participants, regardless of enrollment cohort or dose assignment. As a result, there are no a priori hypotheses for comparing outcomes between dose levels. Of the 42 participants who completed the intervention, n=30 (71.4%) had enough survey data to include in analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (All Participants)
Number analyzed (Participants) | 30
score on a scale | 18.87 (22.49)

4. Secondary Outcome: Within-person Change in Intrinsic Regulation.
Description: This will be assessed using a 4-item measure assessing intrinsic regulation, a subscale of the Behavioral Regulations in Exercise Questionnaire Version 2 (BREQ-2). Items are scored on a 0 (Not true for me) to 4 (Very true for me) scale, and averaged to create a total score, with higher scores indicating greater intrinsic regulation. Pre-specified to report primary and secondary outcome results across the full sample.
Time Frame: Intrinsic regulation (IR) will be assessed at the completion of the 2-week run-in and end of the 2-week follow-up period. Changes in IR will be reported comparing mean difference scores between run-in and follow-up (follow-up mean minus run-in mean)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 30
score on a scale | 0.292 (0.905)

5. Secondary Outcome: Within-person Change in Discrepancy in Behavior.
Description: This will be assessed with a single item measuring discrepancy in behavior. The text of the measure is "How large is the difference between your current walking behavior and your goal concerning your walking?" The question is rated from 1 (Not at all different) to 7 (very different) with higher scores indicating greater levels of discrepancy in behavior. Pre-specified to report primary and secondary outcome results across the full sample.
Time Frame: Discrepancy in behavior (DIB) will be assessed at the completion of the 2-week run-in and end of the 2-week follow-up period. Changes in DIB will be reported comparing mean difference scores between run-in and follow-up (follow-up mean minus run-in mean)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 30
score on a scale | -1.13 (1.36)

6. Secondary Outcome: Within-person Change in Motivation.
Description: Motivation will be assessed with a message stating "I feel motivated to walk each day." Participants will rate this item on a scale of 1 (Not true at all) to 7 (Very true) with higher scores indicating higher levels of motivation. Pre-specified to report primary and secondary outcome results across the full sample.
Time Frame: Motivation will be assessed at the completion of the 2-week run-in and at the end of the 2-week follow-up period. Changes in motivation will be reported comparing the mean difference scores between run-in and follow-up (follow-up mean minus run-in mean)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 30
score on a scale | 0.167 (1.556)

7. Secondary Outcome: Within-person Change in Environmental Context and Resources.
Description: This will be assessed using a checklist of 7 potential barriers to walking. Barriers are coded on a 1 (Not often at all) to 5 (Very often) scale, and averaged to create a total score, with higher scores indicating that the listed barriers had greater effects on walking. Pre-specified to report primary and secondary outcome results across the full sample.
Time Frame: Environmental context and resources (ECaR) will be assessed at completion of 2-week run-in & end of 2-week follow-up period. Changes in ECaR will be reported comparing mean difference scores between run-in & follow-up (follow-up mean minus run-in mean)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 30
score on a scale | 0.176 (0.493)

8. Secondary Outcome: Within-person Change in Medication Adherence.
Description: Participant adherence to statin medication will be assessed continuously using a smart electronic pill bottle. Daily medication adherence will be recorded for each participant across the full duration of the study. Changes in medication between run-in and intervention phases will be compared using Generalized Linear Mixed Model Analyses. Adherence during run-in and follow-up periods will be reported as the proportion of days adherent (e.g. 0.786 for 11 out of 14 days adherent). Changes in adherence between run-in and follow-up will be reported as the mean change in proportion of days adherent
Time Frame: Medication adherence will be assessed continuously via a smart pill bottle and adherence will be calculated daily. Change over time will be examined between the 2-week run-in and the follow-up period (2 weeks post-variable intervention of 5-10 weeks).
Population: Results presented for the full sample. This is an adaptive trial using the TiTE-CRM. Doses are assigned using adaptive methods throughout the trial using all available data from all participants, regardless of enrollment cohort or dose assignment. As a result, there are no a priori hypotheses for comparing outcomes between dose levels. Missing data were treated as non-adherence. Of 42 participants who completed the intervention, all (100%) were analyzed for within-person changes in adherence.
Measure: Mean (Standard Deviation); unit: proportion of medication adherence
Arm/Group | Intervention
Number analyzed (Participants) | 42
proportion of medication adherence | -0.16 (0.29)

9. Other Pre Specified Outcome: Between-person Heterogeneity in Treatment Response.
Description: Participant heterogeneity in amount of time required to reach a successful increase in daily steps (defined as an increase of 2,000 or more steps per day over a 2-week period compared to run-in) will be examined. Average step counts will be calculated for each 2-week block during the intervention and follow-up periods. Average steps per day in these blocks will be compared with the average daily steps in the run-in period. Once a successful increase has been detected, the time to achieve this treatment response will be recorded. Differences in duration to successful increases in physical activity will be examined between participants using mixed effects regression models. Pre-specified to report primary and secondary outcome results across the full sample.
Time Frame: Steps will be assessed continuously via worn activity tracker and step counts will be reported daily. Step counts will be averaged during the 2-weeks of run-in and by 2-week blocks during the intervention and follow-up period (5-14 weeks from run-in).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected across the run-in period (2 weeks pre-intervention), the variable intervention period (5-10 weeks), and the follow-up period (2 weeks post-intervention) for a total of up to 14 weeks.
Arm/Group | Multi-BCT Intervention 5 Weeks | Multi-BCT Intervention 6 Weeks | Multi-BCT Intervention 8 Weeks | Multi-BCT Intervention 9 Weeks | Multi-BCT Intervention 10 Weeks
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/3 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/3 | 0/28
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/3 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05273723/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT05273723/ICF_001.pdf